CLINICAL TRIAL: NCT06042556
Title: A Randomized Trial Evaluating the Effectiveness of a Previously Developed Online IUD Self-removal Guide Versus Basic Information Sheet in Clinical and Non-clinical Settings
Brief Title: IUD Self-Removal: Evaluating an Online Guide for Self-removal in Clinical and Non-clinical Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Kelsey Petrie, Clinical Instructor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00014317
Record Dates: First submitted 2023-09-08; First posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: IUD; Contraception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guide (Experimental): Randomized to use of our IUD self-removal guide
  Interventions: Other: IUD self-removal guide
- No guide (No Intervention): Randomized to use of no additional resource

INTERVENTIONS:
Other: IUD self-removal guide — We previously developed an online guide for IUD self-removal through an iterative process including advice from key expert informants, focus groups, interviews, and a pilot clinical study. It includes an online animation, step-by-step guide, troubleshooting tips, and information about pregnancy and contraception.
  Arms: Guide

SUMMARY:
Investigators previously developed a guide to help people with IUD self-removal. In this randomized study, the goal is to see if this guide makes it easier for IUD-users to remove their own IUDs.

The main question the study aims to answer is:

-Does use of the previously developed IUD self-removal guide increase rates of self removal?

Participants will:

* Complete a pre-study survey
* Be randomized to self-removal with use of the guide or no additional resource
* Self-select participation at home or in clinic
* Attempt IUD self-removal either at home or in clinic
* Complete a post-study survey.

Investigators will compare rates of successful self-removal between those randomized to the guide to those randomized to no additional resource to see if increases success.

ELIGIBILITY:
Inclusion Criteria:

* Ages 14 and older
* IUD in place and desiring removal
* Interest in attempting self-removal
* English speaking
* Working cell-phone with camera.

Exclusion Criteria:

* Not meeting above inclusion criteria, no other specific exclusion criteria

Min Age: 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2021-04-03 (Actual); Primary Completion 2023-02-16 (Actual); Study Completion 2023-02-16 (Actual)

PRIMARY OUTCOMES:
Comparison of successful IUD self-removal rates | The post study survey will be completed within 48 hours of study participation. Participants schedule their participation on average 1-3 months from study enrollment but up to 1 year (the duration of the study being open).
  Successful self-removal will be reported by participants on the post-study survey and documented with an uploaded photo of the removed IUD on a study ruler sheet. Rates of successful self-removal will be compared between those randomized to the guide versus no additional resource.

CONTACTS AND LOCATIONS:
Overall Officials: Kelsey Petrie, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- Cedar River Clinics, Renton, Washington, United States

IPD SHARING:
Plan to Share IPD: No